CLINICAL TRIAL: NCT02814084
Title: Effect of the Prevena Incision Management System on Sternal Wound Edge Perfusion in Patients Undergoing CABG With Bilateral Mammary Artery Grafts
Brief Title: Prevena Incision Management
Acronym: Prevena
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Collaborators: 3M (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STH18497
Record Dates: First submitted 2016-06-08; First posted 2016-06-27 (Estimated); Last update posted 2023-05-24 (Actual); Status verified 2023-05

CONDITIONS: Cardiac Event; Arrest; Cardiac, Complicating Surgery; Coronary Bypass Graft Stenosis; Complication of Coronary Artery Bypass Graft
MeSH Terms: conditions — Cardiovascular Diseases; Heart Arrest

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bilateral Internal Mammary Artery grafts (Active Comparator): Standard care wound dressings used as part of coronary artery bypass graft operation
  Interventions: Device: Bilateral Internal Mammary Artery grafts
- Prevena (Experimental): Prevena dressing used as part of coronary artery bypass graft operation.
  Interventions: Device: Prevena

INTERVENTIONS:
Device: Bilateral Internal Mammary Artery grafts — Sternal Wound Edge Oxygenation in patients undergoing Coronary Artery bypass surgery with Bilateral Internal Mammary Artery grafts
  Arms: Bilateral Internal Mammary Artery grafts
Device: Prevena — The Prevena wound management system applies negative pressure to the closed wound for up to 7 days and is associated with lower rates of surgical site infection.
  Arms: Prevena

SUMMARY:
The question this research project wants to explore is whether using the Prevena Incision Management System (Prevena) will improve sternal wound edge oxygenation in patients undergoing Coronary Artery bypass surgery with Bilateral Internal Mammary Artery grafts.

DETAILED DESCRIPTION:
Coronary artery bypass is the gold standard surgical treatment of patients with complex coronary disease. It is a common operation and more than 16000 procedures per year are carried out in the UK. Recent publications suggest that during the bypass procedure both left and right internal mammary arteries should be used to bypass coronary stenoses. It was noted that using both internal mammary arteries will result in even better long term survival with improved freedom from cardiac events such as myocardial infarction or further coronary intervention than using. The major drawback of using both internal mammary arteries is the increased risk of sternal wound infection and breakdown. The investigators will use Near Infra-Red Spectroscopy (NIRS) to assess the wound edge oxygenation delivery. The NIRS INVOS system the investigators use within Sheffield Teaching Hospitals can measure oxygenation of soft tissue to a certain depth making it suitable for the assessment of wound edge oxygen delivery. Prevena is commercially available and has a CE mark.

The Prevena wound management system differs from conventional wound dressings, it applies negative pressure to the closed wound for 7 days. Wound complications/infections are decreased when this type of wound management system is used. Studies suggest that Prevena achieves these outcomes because of an increase of perfusion in the wound edges and keeping the wound dry. Patients will be randomised to either the Prevena wound management or their standard of care NHS wound management for their procedure. The oxygenation and outcomes of the wounds will be compared through data collection and the patients followed up during their routine inpatient care and 6 week outpatient appointment.

ELIGIBILITY:
Inclusion Criteria:

* Eligible patients are those who require isolated coronary artery bypass surgery, who need at least 2 bypass grafts, and who are deemed suitable by the operating surgeon to have both right and left internal mammary arteries harvested as conduits

Exclusion Criteria:

* Require additional procedures in addition to the coronary bypass or need for internal mammary artery harvest for feasibility study
* Who are deemed by the operating surgeon as unsuitable for bilateral internal mammary artery harvest because of
* Age (75 or older where prognostic benefit of using both internal mammary arteries has been questioned),
* Obesity with a BMI which is higher than 35 (increased risks of wound infection)
* Diabetes (of any type) (increased risks of infection.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2016-09-13 (Actual); Primary Completion 2020-02-09 (Actual); Study Completion 2020-02-09 (Actual)

PRIMARY OUTCOMES:
NIRS measurement of the inferior third of the parasternal region and left forearm assessment | Measurements taken up to 6 weeks post sternotomy wound dressing
  NIRS assessment of the left forearm will also be performed at the same time acting as a control to take into account factors other than wound perfusion that influence oxygen delivery. The difference of the two readings will be the final measurement used for comparison.

SECONDARY OUTCOMES:
Wounds will be scored according to the ASEPSIS scoring system | On the day of dressing removal and at the 6 week postoperative outpatient visit.
  This will be done by an observer who is blinded to the dressing used.

CONTACTS AND LOCATIONS:
Overall Officials: Norman Briffa, Principal Investigator — Sheffield Teaching Hospitals NHS Foundation Trust
Locations (1):
- Sheffield Teaching Hospitals NHS FT, Sheffield, England, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Holmes C, Briffa N. Patient-Reported Outcome Measures (PROMS) in patients undergoing heart valve surgery: why should we measure them and which instruments should we use? Open Heart. 2016 May 5;3(1):e000315. doi: 10.1136/openhrt-2015-000315. eCollection 2016. PMID 27175284
- [Result] Rowe R, Iqbal J, Murali-Krishnan R, Sultan A, Orme R, Briffa N, Denvir M, Gunn J. Role of frailty assessment in patients undergoing cardiac interventions. Open Heart. 2014 Feb 1;1(1):e000033. doi: 10.1136/openhrt-2013-000033. eCollection 2014. PMID 25332792
- [Result] Briffa N. Surgeons' attitudes to intraoperative death. Cardiac surgeons might have different attitudes. BMJ. 2001 Aug 11;323(7308):341-2. No abstract available. PMID 11548680
- [Result] Solodkyy A, Shalhoub J, Chetty G, Briffa NP. A rare case of giant coronary artery aneurysm in the context of multiple arterial aneurysms. Int J Surg Case Rep. 2012;3(7):311-3. doi: 10.1016/j.ijscr.2012.03.023. Epub 2012 Mar 29. PMID 22543232
- [Derived] Jenkins S, Komber M, Mattam K, Briffa N. Negative pressure wound therapy in patients with diabetes undergoing left internal thoracic artery harvest: A randomized control trial. J Thorac Cardiovasc Surg. 2024 Jan;167(1):256-268. doi: 10.1016/j.jtcvs.2022.01.060. Epub 2022 Apr 9. PMID 35550716